CLINICAL TRIAL: NCT03514238
Title: The Irisin and Metabolic Exercise Training Study
Acronym: iMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: New Brunswick Health Research Foundation (Other)
Responsible Party: Principal Investigator, Martin Senechal, Assistant Professor, University of New Brunswick
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: University of New Brunswick
Record Dates: First submitted 2018-04-18; First posted 2018-05-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: Exercise; Physical Activity; Cardio-metabolic Health; Myokines; Cardiorespiratory Fitness; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Motor Activity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults (BMI: ≥30 kg/m2) (Experimental): Obese individuals will participate to three conditions:
  Control Sitting Condition (C), Sitting for 35 minutes Acute Bout of Continuous Moderate Aerobic Exercise (MOD) 50-55% of heart rate reserve Acute Bout of High Intensity Interval Aerobic Exercise (HIIT) 85-90% heart rate reserve
  Interventions: Behavioral: High Intensity Interval Aerobic Exercise (HIIT); Behavioral: Continuous Moderate Aerobic Exercise (MOD); Behavioral: Control Sitting Condition (C)
- Adults (BMI: 18.5-24.9 kg/m2) (Experimental): Normal weight individuals will participate to three conditions:
  Control Sitting Condition (C), Sitting for 35 minutes Acute Bout of Continuous Moderate Aerobic Exercise (MOD) 50-55% of heart rate reserve Acute Bout of High Intensity Interval Aerobic Exercise (HIIT) 85-90% heart rate reserve
  Interventions: Behavioral: High Intensity Interval Aerobic Exercise (HIIT); Behavioral: Continuous Moderate Aerobic Exercise (MOD); Behavioral: Control Sitting Condition (C)

INTERVENTIONS:
Behavioral: High Intensity Interval Aerobic Exercise (HIIT) — Cycling at 50-55% heart rate reserve for 5 minutes followed by 2 minutes of cycling at 85-90% heart rate reserve consecutively for a total of 35 minutes.
  Blood draws will occur at 6 different time points during exercise (0min, 7min, 14min, 21min, 28min, 35min).
Behavioral: Continuous Moderate Aerobic Exercise (MOD) — 35 minutes of cycling at 50-55% heart rate reserve. Blood draws will occur at 6 different time points during exercise (0min, 7min, 14min, 21min, 28min, 35min).
Behavioral: Control Sitting Condition (C) — Blood draws matched for exercise time will be taken while participant remains seated for 35 minutes (0min, 7min, 14min, 21min, 28min, 35min).

SUMMARY:
It has been established that greater amounts of vigorous intensity physical activity lead to improved health outcomes. Interestingly, the response of biologically active substances, called myokines, differs according to exercise intensity. As such, the current study aims to compare the difference in the response to irisin according to different exercise intensities in both normal weight subjects and individuals living with obesity. This study will compare continuous moderate intensity physical activity to high intensity physical activity against a control condition. Furthermore, this study will determine whether differences in exercise intensity are associated with better insulin sensitivity.

DETAILED DESCRIPTION:
Although exercise is recognized as a cornerstone in the management of obesity and diabetes, previous research has shown substantial inter-individual variability following an exercise intervention. As of now, the mechanisms underlying the cardio-metabolic response to exercise have not been fully elucidated. When accounting for genetic factors, only 20-30% of the response is explained, which indicates that other factors must contribute to this exercise-related cardio-metabolic response. Exercise stimulates the release of myokines, which have been shown to play a critical role in health. However, the contribution of these myokines to the cardio-metabolic response is unknown. Furthermore, the regulation of myokines according to different exercise stimuli (i.e., exercise intensity) is unclear. It is suggested that altering specific exercise parameters can reduce the variability in the response and increase the proportion of participants who obtain the expected physiological adaptations.

The purpose of this project is to: 1) determine whether high intensity interval training (HIIT) generates a greater secretion of irisin compared to moderate (MOD) aerobic exercise in individuals living with obesity and in those with a normal weight; 2) investigate whether the increase in irisin during exercise is associated with insulin sensitivity in individuals living with obesity and in those with normal weight; and 3) determine whether differences exist between groups.

Methods: The investigators will use a randomized controlled crossover design to perform this study in which 40 participants (aged 19-50) will be recruited into two groups (n = 20 obese, n = 20 normal weight). Each group will be randomized into three conditions: 1) an acute bout of MOD aerobic exercise: 35 minutes of cycling at 50% of heart rate reserve (HRR), 2) an acute bout of HIIT aerobic exercise: cycling at 50% of HRR for 5 minutes followed by 2 minutes of cycling at 85-90% of HRR consecutively for a total of 35 minutes, and 3) a control condition: blood draws matched for exercise time will be taken while the participant remains seated. The primary outcome measure will be insulin sensitivity using the Matsuda Index. The primary exposure variable will be the acute secretion of irisin during exercise.

Study hypothesis: It is hypothesized that: 1) an acute bout of HIIT aerobic exercise will generate a greater plasma irisin secretion compared an acute bout of continuous MOD aerobic exercise; 2) increased irisin will be positively associated with greater insulin sensitivity; and 3) differences will be observed between individuals living with obesity and those with a normal weight.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (≥30 kg/m2);
* Physical inactivity (must not reach Canadian Physical Activity Guidelines);
* At risk for Type 2 diabetes;
* Adult (aged 19-50).

Exclusion Criteria:

* Individuals with Type 2 diabetes;
* Chronic conditions or injuries that would impact exercise;
* Regular exercise training.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | Baseline
  Insulin sensitivity using the Matsuda Index.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sénéchal, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick - Kinesiology, Fredericton, New Brunswick, Canada

REFERENCES:
- [Background] Fox J, Rioux BV, Goulet EDB, Johanssen NM, Swift DL, Bouchard DR, Loewen H, Senechal M. Effect of an acute exercise bout on immediate post-exercise irisin concentration in adults: A meta-analysis. Scand J Med Sci Sports. 2018 Jan;28(1):16-28. doi: 10.1111/sms.12904. Epub 2017 May 24. PMID 28453881
- [Background] Blizzard LeBlanc DR, Rioux BV, Pelech C, Moffatt TL, Kimber DE, Duhamel TA, Dolinsky VW, McGavock JM, Senechal M. Exercise-induced irisin release as a determinant of the metabolic response to exercise training in obese youth: the EXIT trial. Physiol Rep. 2017 Dec;5(23):e13539. doi: 10.14814/phy2.13539. PMID 29208692
- [Derived] Rioux B, Paudel Y, Thomson A, Peskett L, Senechal M. An examination of exercise intensity and its impact on the acute release of irisin across obesity status: a randomized controlled crossover trial. Appl Physiol Nutr Metab. 2024 Dec 1;49(12):1712-1728. doi: 10.1139/apnm-2024-0091. Epub 2024 Sep 3. PMID 39226615